CLINICAL TRIAL: NCT03145207
Title: Evaluation of Bioavailability of Lidocaine Dermal Products
Brief Title: PK and DPK of Lidocaine Dermal Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HP-00067033
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Heat Effect
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- name brand patch (Other): name brand lidocaine patch
  Interventions: Drug: Lidocaine patch
- generic patch (Other): generic lidocaine patch
  Interventions: Drug: Lidocaine patch
- name brand patch-early (Other): name brand lidocaine patch-early
  Interventions: Drug: Lidocaine patch
- name brand patch-late (Other): name brand lidocaine patch-late
  Interventions: Drug: Lidocaine patch
- generic patch-early (Other): generic lidocaine patch-early
  Interventions: Drug: Lidocaine patch
- generic patch-late (Other): generic lidocaine patch-late
  Interventions: Drug: Lidocaine patch
- both patches (Other): brand name and generic lidocaine patch
  Interventions: Drug: Lidocaine patch

INTERVENTIONS:
Drug: Lidocaine patch — lidocaine patch
  Other Names: skin patch

SUMMARY:
This is a bioequivalence study to compare lidocaine release between a brand name and generic skin patches in healthy adults.

DETAILED DESCRIPTION:
This research study is intended to determine the effect of heat on lidocaine patches. This study will use lidocaine patches (brand name and generic patches) that have been approved by the Food and Drug Administration (FDA) and are already sold to customers in the United States, and will not include any placebos.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant, women who are of any ethnic background between the age of 18 and 45 years old.
2. Subjects must be non-smokers (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches or electronic cigarettes) over the previous 2 months and are not currently using tobacco products.
3. Provide written informed consent before initiation of any of the study procedures.
4. Agrees not to participate in another clinical trial/study or to participate in an investigational drug study for at least 1 month after the last study session.
5. Able to adhere to the study restrictions and protocol schedule.
6. Able to participate in all study sessions.
7. Has a volar forearm of either at least 24 cm (9.45 inches) in length or of sufficient size that can accommodate the formulations to be tested in a study area that begins at least 5 cm (1.97 inches) above the wrist and ends a minimum of 0.5 cm (0.197 inches) below the antecubital fossa (i.e., the bend in the arm at the elbow).
8. Subjects have upper arms (minimum 28 cm (11 inch) circumference) large enough to allow for the placement of two 140 cm2 patches on one upper arm or one 140 cm2 patch on each upper arm.
9. Subjects deemed to be healthy as judged by the MAI and determined by medical history, physical examination and medication history.
10. Negative urine drug screening test.
11. Have normal screening laboratories for WBC, CBC, Hgb, platelets, sodium, potassium, chloride, bicarbonate, BUN, creatinine, ALT and AST.
12. Have normal screening laboratories for urine protein and urine glucose.
13. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e., history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of each procedure day, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner.
14. Agrees not to donate blood to a blood bank throughout participation in the study and at least 3 months after the last procedure day.
15. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute).
16. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-140 mmHg
    * Diastolic blood pressure 60-90 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-20 breaths per minute

Exclusion Criteria:

1. Women who are pregnant, lactating, breast feeding or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of each study session.
2. Smokers (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches or electronic cigarettes).
3. Participation in any ongoing investigational drug trial/study or clinical drug trial/study.
4. History of chronic obstructive pulmonary disease or cor pulmonale, or substantially decreased respiratory reserve, hypoxia, hypercapnia or pre-existing respiratory depression.
5. Active positive Hepatitis B, C and/or HIV serologies (see Appendix B).
6. Known anemia.
7. Positive urine drug screening test.
8. Use of chronic prescription medication during the period 0 to 30 days; or over-the counter medication (e.g. antihistamines or topical corticosteroids) and short term (<30 days) prescription medications during the period 0 to 3 days before a study session (vitamin, herbal supplements and birth control medications not included).
9. Donation or loss of greater than one pint of blood within 60 days of entry to the study.
10. Any prior adverse reaction to lidocaine. Hypersensitivity to lidocaine, known history of hypersensitivity to local anesthetics of the amide type, other excipients in the patches tested or to adhesives on tapes used to cover or tape strip treatment sites.
11. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study.
12. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
13. Consumption of alcohol within 24 h prior to dose administration.
14. History as either reported by the subject or evident to the investigator of infectious disease or skin infection or of chronic skin disease (e.g., diabetes, psoriasis, atopic dermatitis).
15. Hereditary skin disorders or any skin inflammatory conditions as reported by the research participant or evident to the MAI.
16. History of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and did not involve the investigative sites.
17. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at application site (volar forearms/upper arms), sunburn, raised moles and scars, open sores at application site (volar forearms/upper arms), scar tissue, tattoo or coloration that would interfere with placement of formulations, skin assessment or reactions to lidocaine.
18. BMI ≥30 kg/m2.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra Stinchcomb, PhD, Principal Investigator — University of Maryland Baltimore School of Pharmacy; Hazem Hassan, PhD, Principal Investigator — University of Maryland Baltimore School of Pharmacy
Locations (1):
- General Clinical Research Center (GCRC) at the University of, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine: Session 1-name brand patch Session 2-generic lidocaine patch Session 3-name brand patch with early heat application Session 4-name brand patch with late heat application Session 5-generic patch with early heat application Session 6-generic patch with late heat application Session 7-name brand and generic lidocaine patch pieces with skin tape stripping
  The same 12 volunteers completed each of the seven study sessions.
Period: Overall Study
Arm/Group | Lidocaine
Started | 14 (The same 12 volunteers completed each of the seven study sessions.)
Completed | 12
Not Completed | 2
Not completed — volunteer started taking allergy shots | 1
Not completed — baseline blood pressure high | 1

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine: Session 1-name brand patch Session 2-generic lidocaine patch Session 3-name brand patch with early heat application Session 4-name brand patch with late heat application Session 5-generic patch with early heat application Session 6-generic patch with late heat application Session 7-name brand and generic lidocaine patch pieces with skin tape stripping
Arm/Group | Lidocaine
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.14 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Maximum Serum Concentration (Cmax)
Description: maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered
Time Frame: six study sessions for each participant; through 15 h each study session
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lidocaine Name Brand Patch: Session 1-name brand patch
- Lidocaine Generic Patch: Session 2-generic lidocaine patch
- Lidocaine Name Brand Patch Early Heat: Session 3-name brand patch with early heat application
- Lidocaine Name Brand Patch Late Heat: Session 4-name brand patch with late heat application
- Lidocaine Generic Early Heat: Session 5-generic patch with early heat application Session 6-generic patch with late heat application Session 7-name brand and generic lidocaine patch pieces with skin tape stripping
- Lidocaine Generic Late Heat: Session 6-generic patch with late heat application
Arm/Group | Lidocaine Name Brand Patch | Lidocaine Generic Patch | Lidocaine Name Brand Patch Early Heat | Lidocaine Name Brand Patch Late Heat | Lidocaine Generic Early Heat | Lidocaine Generic Late Heat
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
ng/mL | 306.8 (756.3) | 214.9 (280.5) | 390.76 (387.29) | 286.49 (288.59) | 368.09 (348.93) | 314.95 (287.36)

ADVERSE EVENTS:
Time Frame: TL-001 (58 days), TL-003 (113 days), TL-005 (135 days), TL-007 (62 days), TL-010 (72 days), TL-017 (388 days), TL-020 (272 days), TL-022 (693 days), TL-023 (61 days), TL-025 (358 days), TL-030 (97 days), TL-031 (108 days)
Arm/Group | Name Brand Patch | Generic Patch | Name Brand Patch-early | Name Brand Patch-late | Generic Patch-early | Generic Patch-late | Both Patches
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 13/14 | 9/14 | 11/13 | 11/13 | 12/12 | 12/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Name Brand Patch (N=14) | Generic Patch (N=14) | Name Brand Patch-early (N=13) | Name Brand Patch-late (N=13) | Generic Patch-early (N=12) | Generic Patch-late (N=12) | Both Patches (N=12)
headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
decreased heart rate (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
increased respiratory rate (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
decreased blood pressure (General disorders) | 4 (4) | 2 (2) | 5 (5) | 4 (4) | 3 (3) | 6 (6) | 4 (4)
increased blood pressure (General disorders) | 2 (2) | 2 (2) | 0/12 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
skin itching (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
hyperpigmentation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
erythema (General disorders) | 6 (6) | 4 (4) | 6 (6) | 6 (6) | 5 (5) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03145207/Prot_SAP_000.pdf